CLINICAL TRIAL: NCT05783713
Title: Evaluation of the Effectiveness of a Flu Vaccination Campaign for Healthcare Workers of the Fondazione Policlinico Universitario "A. Gemelli" IRCCS and the Catholic University of the Sacred Heart (UCSC): a Pre-post Study
Brief Title: Evaluation of the Effectiveness of a Flu Vaccination Campaign for Healthcare Workers of a Teaching Hospital: a Pre-post Study
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 2263
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Influenza Vaccination
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Influenza Vaccination — Describe and measure any differences in total influenza vaccination coverage, in different categories of professionals and in different operational units.

SUMMARY:
The goal of this observational study is to evaluate the effectiveness of the vaccination strategy implemented during the 2019/2020 flu vaccination campaign compared with the previous one. The main question it aims to answer is whether there are differences in the total coverage of influenza vaccination, in different categories of professionals and in different operating units.

ELIGIBILITY:
Inclusion Criteria:

* Health personnel employed by the Fondazione Policlinico Universitario "A. Gemelli" IRRCS

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health personnel employed by the Fondazione Policlinico Universitario "A. Gemelli" IRRCS
Sampling Method: Non-Probability Sample
Enrollment: 10737 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
influenza vaccination coverage | 16 months
  Describe and measure differences in total influenza vaccination coverage between the vaccination seasons considered, in different categories of professionals and in different operational units.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario "A. Gemelli" IRCCS, Roma, RM, Italy